CLINICAL TRIAL: NCT06542588
Title: A Multicenter, Single-arm, Open-label Clinical Trial of Short-Course Radiotherapy Followed by Neoadjuvant Chemotherapy, HLX07 and Serplulimab in the Treatment for RAS/BRAF Wild Type Locally Advanced Rectal Cancer
Brief Title: Short-Course Radiotherapy Followed by Neoadjuvant Chemotherapy, HLX07and Serplulimab in LARC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX10IIT170
Record Dates: First submitted 2024-08-04; First posted 2024-08-07 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-08

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Short course radiotherapy sequential HLX07, Serplulimab and chemotherapy (Experimental): Radiotherapy will employ conformal or intensity-modulated radiation therapy, with a pelvic irradiation dose of 25 Gy/5 Fractions/1 week. Then rest for 1 week after radiotherapy and begin to receive neoadjuvant chemotherapy CAPOX, HLX07 and Serplulimab, for 6 cycles.
  The patients were operated within 10 weeks after the last treatment, and the surgical method is total mesorectal excision. For patient who achieve CR can choose non-operation management.
  Interventions: Combination Product: HLX07(anti EGFR antibody) and Serplulimab(anti PD-1 antibody)

INTERVENTIONS:
Combination Product: HLX07(anti EGFR antibody) and Serplulimab(anti PD-1 antibody) — Short course radiotherapy sequential HLX07, Serplulimab and chemotherapy
  Other Names: CAPOX

SUMMARY:
The study is a multicenter, open-label, phase II clinical study, and the purpose of the study is to explore the complete response rate (CR, Defined as pathological complete response (pCR) + Clinical complete response (cCR)) of patients with RAS/BRAF wild type locally advanced rectal cancer(LARC) treated with short-term radiotherapy, sequential HLX07, Serplulimab and CAPOX. A total of 29 patients were included in this study.

DETAILED DESCRIPTION:
Patients with RAS/BRAF wild type locally advanced rectal cancer (T3-4/N+) , combined risk factors, will be treated with neoadjuvant therapy, and the Primary endpoint of the study is complete response rate(CR, Defined as pathological complete response (pCR) + Clinical complete response (cCR) ). PCR assessed by the blind independent review committee (BIRC), defined as the absence of viable tumour cells in the resected primary tumour specimen and all sampled regional lymph nodes (ypT0N0). CCR evaluation was based on a combination of digital rectal examination, endoscopy, rectal MRI and blood carcinoembryonic antigen levels.

ELIGIBILITY:
Inclusion Criteria:

1. Patients or their family members agree to participate in the study and sign the informed consent form;
2. Age 18-75 years, male or female;
3. Histologically confirmed Locally Advanced rectal adenocarcinoma
4. Genetic test and/or immunohistochemical confirmation of RAS, BRAF wild type
5. inferior margin ≤ 10 cm from the anal verge;
6. Pelvic MRI shows high risk [meets one of the following conditions]:

   * Clinical tumor (cT) staging cT4a or cT4b (according to AJCC 8th Edition)
   * Extramural vascular infiltration
   * Clinical lymph node (cN) staging cN2 (according to AJCC 8th Edition)
   * Mesenteric fascia is involved
   * Lateral lymph node enlargement 7 ECOG performance status score is 0-1;

8. Swallowing pills normally; 9. Untreated with anti-tumor therapy for rectal cancer, including radiotherapy, chemotherapy, surgery, etc; 10. There was no operative contraindication; 11. Laboratory tests were required to meet the following requirements: white blood cell (WBC) ≥ 4×109/L; Absolute neutrophil count (ANC) ≥ 1.5×109/L; Platelet count ≥ 100×109/L; Hemoglobin ≥90 g/L; Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN); Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN; Serum creatinine ≤1.5 times the upper limit of normal value or creatinine clearance rate ≥50 mL/min; International normalized ratio (INR) ≤ 1.5 × ULN; Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN 12. Males or females with reproductive ability who are willing to use contraception in the trial;

Exclusion Criteria:

1. Documented history of allergy to study drugs, including any component of Anti-EGFR or PD-1 antibody, capecitabine, oxaliplatin and other platinum drugs;
2. Have received or are receiving any of the following treatments:

   Any radiotherapy, chemotherapy or other anti-tumor drugs for tumor; Patients who need to be treated with corticosteroid (dose equivalent to prednisone of >10 mg/day) or other immunosuppressive agents within 2 weeks prior to study drug administration; Received live attenuated vaccine within 4 weeks before the first use of the study drug; Major surgery or severe trauma within 4 weeks before the first use of the study drug;
3. Any active autoimmune disease or history of autoimmune disease;
4. Have a history of immunodeficiency, including HIV positive, or other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation or allogeneic bone marrow transplantation;
5. There are clinical symptoms or diseases of heart that are not well controlled;
6. Severe infection (CTCAE > 2) occurred within 4 weeks before the first use of the study drug; Baseline chest imaging revealed active pulmonary inflammation, signs and symptoms of infection within 14 days prior to the first use of the study drug, or oral or intravenous antibiotic therapy, except for prophylactic use of antibiotics;
7. Patients with active pulmonary tuberculosis infection found by medical history or CT examination, or with a history of active pulmonary tuberculosis infection within one year before enrollment, or with a history of active pulmonary tuberculosis infection more than one year ago but without regular treatment;
8. The presence of active hepatitis B (HBV DNA > 2000 IU/mL or 104 copies/mL) was positive for hepatitis C (hepatitis C antibody) and HCV RNA was higher than the lower limit of analytical method;
9. Female subject who is pregnant or breastfeeding;
10. Patients who are not suitable for participation in clinical trials in the opinion of the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
complete response (CR) rate | an expected average of 12 months
  Defined as pathological complete response (pCR) + Clinical complete response (cCR)

SECONDARY OUTCOMES:
3-year disease-Free Survival | an expected average of 3 years
  The time from the first day of disease free (operation date) to local or distant recurrence, or the death event caused by any reason, whichever occurs first
Overall Survival | an expected average of 5 years
  The time from the date of randomization to the death caused by any cause
dverse events (AEs) were graded according to the NCI CTCAE version 5·0 | an expected average of 1.5 years
  Adverse events and surgical safety

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Lin, MD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (2):
- China (2):
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Hubei